CLINICAL TRIAL: NCT02079038
Title: A Prospective, Multi-center, Randomized Controlled Double-Blind Trial Evaluating the VertiFlex® Totalis™ Direct Decompression System Versus a Sham Comparator Surgical Procedure in Patients With Lumbar Spinal Stenosis
Brief Title: The STEPS - Totalis™ Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VertiFlex, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-TDDS-01
Record Dates: First submitted 2014-02-24; First posted 2014-03-05 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Totalis™ Direct Decompression Procedure (Active Comparator): Totalis
  Interventions: Device: Totalis
- Comparator Procedure (Active Comparator): Comparator Surgical Procedure
  Interventions: Procedure: Comparator Surgical Procedure

INTERVENTIONS:
Device: Totalis
  Arms: Totalis™ Direct Decompression Procedure
Procedure: Comparator Surgical Procedure
  Arms: Comparator Procedure

SUMMARY:
The purpose of this study is to determine safety and effectiveness, as measured by changes in pain, disability, patient satisfaction, and claudicatory symptoms, at 6 months following treatment with the Totalis™ Direct Decompression System or Sham Comparator Surgical Procedure in patients with lumbar spinal stenosis

DETAILED DESCRIPTION:
Subjects suffering from symptoms of neurogenic intermittent claudication secondary to a radiographically-confirmed diagnosis of central canal stenosis, with or without mild or moderate lateral recess stenosis, at one or two levels from L1 to L5 who meet all inclusion/exclusion criteria, including ≥6 months of non-operative management.

Patients included in the clinical investigation will return for follow-up visits at 1 week for safety evaluation, and at 6 weeks, 3 months, 6 months, 12 months, 18 months and 24 months post-treatment to collect data for evaluation of safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects greater than or equal to 55 years of age
* Neurogenic intermittent claudication (NIC) symptoms defined generally as leg/buttock/ groin pain and/or paresthesias that are exacerbated with standing and walking and relieved by flexion
* VAS leg symptom severity >50 (in either leg) during episodes of neurogenic claudication
* Subjects who are able to walk a minimum of 50 feet without experiencing NIC symptoms
* Diagnosis of central canal spinal stenosis, with or without mild to moderate lateral recess stenosis, at one or two levels from L1-L5 with radiologic evidence
* Subjects with persistent lumbar spinal stenosis symptoms that, during the course of the last year, have been unresponsive to a minimum of 6 months of conservative therapy

Exclusion Criteria:

* Significant back, buttock or leg pain from causes other than lumbar central canal stenosis
* Axial back pain only
* Severe foraminal stenosis at index level(s) and/or symptomatic foraminal stenosis at any lumbar level
* Severe lateral recess stenosis
* Lumbar spinal stenosis at more than two levels determined pre-operatively to require surgical intervention
* Prior decompressive surgery at index level (s) or fusion at any lumbar level
* Epidural steroid or nerve block steroid injection at index level(s) within 6 weeks of baseline assessments
* Spondylolisthesis (anterolisthesis or retrolisthesis) greater than grade 1
* Spondylolysis (pars fracture)
* Significant degenerative lumbar scoliosis at index level(s)
* Morbid obesity
* Significant peripheral vascular disease
* Active significant co-morbidity
* Undergoing immunosuppressive therapy or long-term steroid use
* Current spinal cord stimulator or implanted pain pump
* Life expectancy less than 2 years
* Evidence of substance abuse within the year
* Involvement or potential involvement in litigation related to the spine or worker's compensation related to a back and/or leg issue

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Hope Research Institute, Phoenix, Arizona
  - Arizona Pain Specialists, Scottsdale, Arizona
  - Medhat Mikhael, M.D. Inc., Fountain Valley, California
  - Orthopedic Pain Specialists, Santa Monica, California
  - Integrated Pain Management Medical Group, Inc., Walnut Creek, California
  - GWU - Medical Faculty Associates, Inc., Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Pain Institute, Merritt Island, Florida
  - Pain Care, LLC, Stockbridge, Georgia
  - American Health Network, Muncie, Indiana
  - Pain Management Associates, Independence, Missouri
  - University Pain Medicine Center, Somerset, New Jersey
  - Oklahoma Pain Physicians, Oklahoma City, Oklahoma
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Performance Spine and Sports Physicians, PC, Pottstown, Pennsylvania
  - SC Pain & Spine Specialists, Murrells Inlet, South Carolina
  - Spine Team Texas, Southlake, Texas
  - Virginia iSpine Physicians PC, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 180 subjects enrolled; 12 withdrew, leaving 168 subjects randomized & treated.
Groups:
- Totalis: Totalis™ Direct Decompression Procedure
- Control Procedure: Comparator Surgical Procedure
Period: Modified Intent to Treat Population
Arm/Group | Totalis | Control Procedure
Started | 112 | 56
Completed | 105 | 51
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Death | 1 | 0
Period: Completed 6 Months
Arm/Group | Totalis | Control Procedure
Started | 105 | 51
Completed | 103 | 50
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Population
Groups:
- Totalis: Totalis ™ Direct Decompression Procedure
- Total: Total of all reporting groups
Arm/Group | Totalis | Control Procedure | Total
Number analyzed (Participants) | 112 | 56 | 168
Age, Customized [Mean (Standard Deviation); unit: years] | 70.8 (10.4) | 71.8 (7.7) | 71.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 36 | 94
  Male | 54 | 20 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 109 | 54 | 163
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Clinically Significant Improvement in Outcomes
Description: Where clinically significant improvement in outcomes is defined as improvement in any 2 of the 3 domains of the Zurich Claudication Questionnaire ( ZCQ)
  * Improvement in physical function by ≥ 0.5 points from baseline
  * Improvement in symptom severity by ≥ 0.5 points from baseline
  * Patient Satisfaction Score of < 2.5 points
  And no interventions of the following nature through 6 months:
  * Re-operations or revisions at index level(s) intended to treat stenosis
  * Epidural steroid injection or selective nerve root block at index level(s)
  And no unblindings
Time Frame: Baseline and 6 Months
Measure: Number; unit: percentage of subjects
Arm/Group | Totalis | Control Procedure
Number analyzed (Participants) | 103 | 50
percentage of subjects | 56.3 | 56.0

ADVERSE EVENTS:
Time Frame: 6 Months
Description: Serious Adverse Events assessed at study visits from Surgical Procedure Visit to End of Study
Arm/Group | Totalis | Control Procedure
All-Cause Mortality (participants affected / at risk) | 1/112 | 0/56
Serious Adverse Events (participants affected / at risk) | 19/112 | 11/56
Other Adverse Events (participants affected / at risk) | 98/112 | 42/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Totalis (N=112) | Control Procedure (N=56)
Cervical Instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (2) | 1 (1)
Pain - Back and Leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal Carcinoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Total Knee Replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trauma from Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aortic regurgitation (Vascular disorders) | 1 (1) | 0 (0)
Non-alcoholic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Death from atherosclerosis (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 2 (2) | 0 (0)
Dyspnea (Cardiac disorders) | 0 (0) | 1 (1)
Gall stones (Hepatobiliary disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 2 (2)
Pain -- Leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subluxed patella (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain -- Toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Totalis (N=112) | Control Procedure (N=56)
Injury, accidental (Injury, poisoning and procedural complications) | 22 (34) | 10 (16)
Pain -- back (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (7)
Pain -- leg (Musculoskeletal and connective tissue disorders) | 15 (16) | 9 (13)
Pain -- buttocks or groin (Musculoskeletal and connective tissue disorders) | 10 (11) | 2 (3)
Neurologiocal disorder, any (Nervous system disorders) | 10 (17) | 4 (7)
Spinal stenosis symptoms at index level (Musculoskeletal and connective tissue disorders) | 14 (19) | 6 (8)
Urinary tract infection (Renal and urinary disorders) | 8 (12) | 0 (0)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days